CLINICAL TRIAL: NCT01966692
Title: Evaluation of the Sensitivity of Pharmacokinetics to Differences in the Aerodynamic Particle Size Distribution of Three Different Formulations of Fluticasone Propionate Dry Powder Inhalers
Brief Title: Sensitivity of Pharmacokinetics to Differences in Aerodynamic Particle Size Distribution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: IRB201400464-need FDA approval; 00079088 (Other: United States: Food and Drug Adminstration); HHSF223401610099C (Other Grant/Funding Number: US FOOD AND DRUG ADMN); OCR15966 (Other: University of Florida)
Record Dates: First submitted 2013-09-30; First posted 2013-10-21 (Estimated); Results first posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2023-11

CONDITIONS: Asthma
Keywords: Bioequivalence; Fluticasone Propionate
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Fluticasone Propionate Formulation Sequence 1233* (Active Comparator): Patients first received Fluticasone Propionate Drug formulation 1, after a washout period of at least 5 days, they then received Fluticasone Propionate Drug formulation 2, after a washout period of at least 5 days, they then received Fluticasone Propionate Drug formulation 3, after a washout period of at least 5 days, they then received Fluticasone Propionate Drug formulation 3*.
  All Fluticasone Propionate Drug formulations were administered via Plastiape Monodose Dry Powder Inhaler, 500mcg single dose.
  Mass Median Aerodynamic Diameter (MMAD) for formulation 1 is 4.5 µm. MMAD for formulation 2 is 3.8 µm MMAD for formulation 3 is 3.7 µm. MMAD for formulation 3* is 3.7 µm. See Formulation Development in Detailed Description for details regarding differences in formulations
  Interventions: Drug: Fluticasone Propionate Formulation 1; Drug: Fluticasone Propionate Formulation 2; Drug: Fluticasone Propionate Formulation 3; Drug: Fluticasone Propionate Formulation 3*
- Fluticasone Propionate Formulation Sequence 23*13 (Active Comparator): Patients first received Fluticasone Propionate Drug formulation 2, after a washout period of at least 5 days, they then received Fluticasone Propionate Drug formulation 3*, after a washout period of at least 5 days, they then received Fluticasone Propionate Drug formulation 1, after a washout period of at least 5 days, they then received Fluticasone Propionate Drug formulation 3.
  All Fluticasone Propionate Drug formulations were administered via Plastiape Monodose Dry powder Inhaler, 500mcg single dose.
  MMAD for formulation 1 is 4.5 µm. MMAD for formulation 2 is 3.8 µm. MMAD for formulation 3 is 3.7 µm. MMAD for formulation 3* is 3.7 µm. See Formulation Development in Detailed Description for details regarding differences in formulations
  Interventions: Drug: Fluticasone Propionate Formulation 1; Drug: Fluticasone Propionate Formulation 2; Drug: Fluticasone Propionate Formulation 3; Drug: Fluticasone Propionate Formulation 3*
- Fluticasone Propionate Formulation Sequence 313*2 (Active Comparator): Patients first received Fluticasone Propionate Drug formulation 3, after a washout period of at least 5 days, they then received Fluticasone Propionate Drug formulation 1, after a washout period of at least 5 days, they then received Fluticasone Propionate Drug formulation 3*, after a washout period of at least 5 days, they then received Fluticasone Propionate Drug formulation 2.
  All Fluticasone Propionate Drug formulations were administered via Plastiape Monodose Dry Powder Inhaler, 500mcg single dose.
  MMAD for formulation 1 is 4.5 µm. MMAD for formulation 2 is 3.8 µm MMAD for formulation 3 is 3.7 µm. MMAD for formulation 3* is 3.7 µm. See Formulation Development in Detailed Description for details regarding differences in formulations
  Interventions: Drug: Fluticasone Propionate Formulation 1; Drug: Fluticasone Propionate Formulation 2; Drug: Fluticasone Propionate Formulation 3; Drug: Fluticasone Propionate Formulation 3*
- Fluticasone Propionate Formulation Sequenct 3*321 (Active Comparator): Patients first received Fluticasone Propionate Drug formulation 3*, after a washout period of at least 5 days, they then received Fluticasone Propionate Drug formulation 3, after a washout period of at least 5 days, they then received Fluticasone Propionate Drug formulation 2, after a washout period of at least 5 days, they then received Fluticasone Propionate Drug formulation 1.
  All Fluticasone Propionate Drug formulations were administered via Plastiape Monodose Dry powder Inhaler, 500mcg single dose. * (The asterisk) A different set of capsules from the same batch of formulation 3 is given to the subject to assess the within-subject variability and to ensure that the study is sufficiently powered to show bioequivalence between two replicates of the same formulation.
  MMAD for formulation 1 is 4.5 µm. MMAD for formulation 2 is 3.8 µm MMAD for formulation 3 is 3.7 µm. MMAD for formulation 3* is 3.7 µm.
  Interventions: Drug: Fluticasone Propionate Formulation 1; Drug: Fluticasone Propionate Formulation 2; Drug: Fluticasone Propionate Formulation 3; Drug: Fluticasone Propionate Formulation 3*

INTERVENTIONS:
Drug: Fluticasone Propionate Formulation 1 — Fluticasone Propionate dry powder inhaler Formulation 1
Drug: Fluticasone Propionate Formulation 2 — Fluticasone Propionate dry powder inhaler Formulation 2
Drug: Fluticasone Propionate Formulation 3 — Fluticasone Propionate dry powder inhaler Formulation 3
Drug: Fluticasone Propionate Formulation 3* — Fluticasone Propionate dry powder inhaler Formulation 3*
  *(The asterisk) A different set of capsules from the same batch of formulation 3 is given to the subject to assess the within-subject variability and to ensure that the study is sufficiently powered to show bioequivalence between two replicates of the same formulation.

SUMMARY:
When a drug company first develops a drug, the company has to show the Food and Drug Administration (FDA) that the drug is safe and effective. If FDA concludes that the drug is safe and effective, FDA approves the drug. The company can then sell the drug, which the company does using "trade name." Only the drug company that developed the "trade name" drug is allowed to sell it. However, other drug companies can create their own version of the "trade name" drug, which usually happens after the patents for the "trade name" product run out. These drugs, often called "generic drugs," potentially will be less expensive for the patient. In order to sell generic drugs, drug companies must show that their generic version is the same as the "trade name" drug in a number of ways. For example, they generally have to show that their product is intended to be used to treat the same diseases or conditions, that it has the same label, and that the product has the same active ingredient as the "trade name" drug. The generic company also has to show that generic product is "bioequivalent" to the trade name drug, meaning that the generic product gets to the part of the body where the drug works at the same rate that the trade name drug does. How to show how much drug gets to the part of the body where it works, and how fast, depends on the type of product the drug is. The primary aim of this research study is to aid the FDA in finding methods to ensure that the versions of generic drugs that are inhaled (for example, drugs used to treat asthma) are bioequivalent to the trade name drug. As a part of the research study, pharmacokinetic (PK) studies (studies measuring drug levels in the blood over time after inhalation) will be done using three different versions of fluticasone propionate (FP, a drug routinely used in asthmatic patients) administered using a dry powder inhaler (DPI, an inhalation device that delivers the drug as a dry powder). The results from this study will help FDA ensure that generic products are the same as the trade name drugs.

DETAILED DESCRIPTION:
Formulation Development

The aim of the pharmaceutical development was to manufacture three Dry powder Inhalation (DPI) formulations containing Fluticasone Propionate in an Plastiape Monodose DPI device, which provide distinct in vitro deposition patterns on a Next Generation Impactor. NGI is a high performance cascade impactor used to characterize aerosol particles by particle size. It is desirable to develop three formulations with the same emitted dose (ED), impactor size mass (ISM) but different mass median aerodynamic diameter (MMAD). Meeting these design criteria for the formulations would help to see if pharmacokinetic parameters are sensitive to regional differences in drug deposition whilst having the dose deposited in the lung from different formulations being the same.The three formulation developed are labeled Fluticasone Propionate Drug formulation 1 through 3.

Study Procedures and scheduling

The study is comprised of 5 visits in total - a screening visit and 4 treatment visits. At least 5 days should lapse between the treatment visits.

Screening Visit During the screening visit, the inclusion and exclusion criteria will be reviewed to ensure the volunteer is appropriate for the study. The informed consent will be reviewed with the volunteer by a member of the study team and the volunteer will be encouraged to ask questions to ensure the volunteer has a good understanding of the study. If the volunteer is eligible and agrees to participate, the volunteer will be asked to sign the informed consent form prior to any study specific procedures including randomization. After the volunteer signs the informed consent, the volunteer will be interviewed and demographic data, medical history and concomitant medications will be collected and recorded. A physical examination will be performed after the vital sign measurements are obtained. A pregnancy test for female volunteers will be obtained. Spirometry testing and inhalation training will be performed by a qualified study clinician/investigator to ensure the suitability of volunteers. Laboratory tests including a Complete Blood Count (CBC), urinalysis and metabolic panel will be collected via venipuncture and processed in the lab. Screening tests will be performed within 14 days of treatment visit 1 and no later than 2 days before treatment visit 1. All screening results will be evaluated by the study clinician/investigator against the inclusion/exclusion criteria to confirm the eligibility of the volunteers.

Inhalation training: Inhalation training will be performed by a qualified study clinician at the screening visit and at each study visit. The training will be accomplished by instructions and subsequent inhalation via training devices containing empty capsules. The instructions on how to use the device correctly are similar to the Foradil Aerolizer DPI product information label. (http://www.rxlist.com/foradil-drug/medication-guide.htm )

Treatment Visits 1, 2, 3 and 4 Eligible volunteers will be asked to return for treatment visit 1. A minimum period of 5 days should lapse between the subsequent treatment visits. Each treatment visit is scheduled for 28 hours over two days. The study will be conducted at the University of Florida (UF) CRC (Clinical Research Center). It is an outpatient study and the volunteer will be asked to come back the following day for the 24 hour blood sample. The volunteer will be asked to stay in an outpatient room during the treatment visit. The same activities are carried out at the other treatment visits.

At each treatment visit, eligibility criteria will be reviewed and confirmed to ensure volunteer is appropriate for study. Changes in medical history including concomitant medications will be documented. Vital signs will be obtained. Inhalation training will be provided to the volunteers as mentioned in the section above. An IV catheter will be inserted in a vein located in the forearm region of the volunteer. The IV catheter is used to avoid multiple pricks while collecting blood samples. The IV catheter is not used for the administration of the drug. The volunteer inhales 5 times from a given inhaler during each treatment visit. Each inhaler will be used only once and by only one volunteer to ensure the volunteer's safety from infectious agents. The schedule below summarizes the procedures performed at the screening visit and a single treatment visit.

Blood sample collection Blood samples will be drawn by inserting an indwelling catheter into the volunteer's median cubital vein in the forearm region. Blood samples will be taken 15 minutes prior to the dosing of the product (pre-dose sample) and 5, 10, 15, 20, 30, 45, 60 minutes, 1.5, 2, 3, 4, 6, 8, 10, 12, 14 and 24 hours post dosing. At each time point 9ml of blood sample will be collected of which the first 1ml will be discarded and the remaining 8 ml will be stored in a vacutainer tube for plasma preparation and storage.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects aged 18 to 50 years (inclusive).
2. Females will be eligible only if they are currently non-lactating and demonstrate a negative urine pregnancy test. Female subjects must be willing to use highly effective methods of contraception throughout the study. A highly effective method of birth control is defined as one which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly e.g. no sexual intercourse, an intrauterine device (IUD), using contraceptive foam AND a condom (double-barrier).
3. Body weight ranging from 50 to 100 kg, corresponding to a BMI of 18-29 kg/m2.
4. Non-smoker for at least 12 months prior to study screening and a maximum smoking history of less than ten-pack years (i.e. the equivalent of one-pack per day for ten years).
5. Healthy and free of significant abnormal findings as determined by medical history, physical examination, vital signs, laboratory tests (including serum cortisol at screening), complete blood count (CBC) with differential, urinalysis and basic metabolic panel.
6. Ability to read, comprehend and sign the consent form.
7. Ability and willingness to comply with all study procedures, discontinue and/or withhold medications as specified in the protocol, and attend scheduled study visits.
8. No history of respiratory disease.
9. Normal baseline spirometry as predicted for age, sex and height, including forced expiratory volume in 1 second / forced vital capacity (FEV1/FVC) > 0.8.
10. Healthy and without any pre-existing medical conditions.

Exclusion Criteria:

1. Any history and/or conditions that might interfere with drug absorption, distribution, metabolism or excretion of FP, e.g., pre-existing lung and liver disease.
2. Known or suspected sensitivity to Flonase (Fluticasone Propionate), Veramyst (Fluticasone Furoate), or related compounds in that class.
3. Hypersensitivity to milk proteins or lactose (inactive ingredients in the formulation).
4. Having a history and/or currently having the medical condition in the opinion of medically accountable investigator and hence taking any medication for the following (including but not limited to):

   4.1 Significant cardiac, dermatologic, gastrointestinal, hepatic, renal, hematological, neurological and psychiatric disease (determined by physical exam, CBC with differential, urinalysis, basic metabolic panel and medical history).

   4.2 Presence of glaucoma, cataracts, ocular herpes simplex or carcinoma (other than basal cell).

   4.3 Presence of tuberculosis and other respiratory diseases (including but not limited to intermittent or persistent asthma, emphysema and chronic bronchitis); or respiratory infection, common cold, sinusitis or ear infections.
5. Current use of hormone replacement therapy (HRT), hormonal contraceptives and/or corticosteroid treatment within the last 2 months.
6. Smoker during the last 1 year prior to study screening (self-report).
7. Evidence of a positive pregnancy urine test for female volunteers or females who are pregnant or breast-feeding or are likely to become pregnant during the trial. Women of child-bearing potential may be included in the study if, in the opinion of the investigator, they are taking adequate contraceptive precautions as described above.
8. Exposure to any investigational drug within 30 days of enrolment.
9. Subjects who are unable to demonstrate proper inhalation of the test products.
10. Subjects who have a history of anemia.
11. Exposure to any medication that alters CYP3A4 activity within last 2 weeks (e.g.: azole antifungals, rifampin).
12. Nausea, vomiting or diarrhoea within 7 days of dosing.
13. Subjects who have donated 1 pint (450 mL) of blood or more within the previous 8 weeks prior to study administration.
14. Any history or current drug or alcohol abuse, which would interfere with the subject's completion of the study and with adherence to the protocol.
15. A subject will not be eligible for this study if he/she is an immediate family member of the participating investigator, sub-investigator, study coordinator, or employee of the participating investigator.
16. The subject is the student of the Principal Investigator (PI).
17. Lack of willingness to have personal study related data collected, archived and transmitted according to the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-01-20 (Actual); Study Completion 2018-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Bulitta, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Sharing of subject's de-identified data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 17 participants screen failed. Total number of participants enrolled into the study was 24.
Groups:
- Fluticasone Propionate Formulation Sequence 1233*: Fluticasone Propionate Drug formulation 1 (500mcg single dose, 1 day), at least 5 days washout, Fluticasone Propionate Drug formulation 2 (500mcg single dose, 1 day), at least 5 days washout, Fluticasone Propionate Drug formulation 3 (500mcg single dose, 1 day), at least 5 days washout, Fluticasone Propionate Drug formulation 3* (500mcg single dose, 1 day)
  See Formulation Development in Detailed Description for details regarding differences in formulations.
  *(The asterisk) A different set of capsules from the same batch of formulation 3 is given to the subject to assess the within-subject variability and to ensure that the study is sufficiently powered to show bioequivalence between two replicates of the same formulation.
- Fluticasone Propionate Formulation Sequence 23*13: Fluticasone Propionate Formulation Sequence 23*13
  Fluticasone Propionate Drug formulation 2 (500mcg single dose, 1 day), at least 5 days washout, Fluticasone Propionate Drug formulation 3* (500mcg single dose, 1 day), at least 5 days washout, Fluticasone Propionate Drug formulation 1 (500mcg single dose, 1 day), at least 5 days washout, Fluticasone Propionate Drug formulation 3 (500mcg single dose, 1 day)
  See Formulation Development in Detailed Description for details regarding differences in formulations.
  *(The asterisk) A different set of capsules from the same batch of formulation 3 is given to the subject to assess the within-subject variability and to ensure that the study is sufficiently powered to show bioequivalence between two replicates of the same formulation.
- Fluticasone Propionate Formulation Sequence 313*2: Fluticasone Propionate Drug formulation 3 (500mcg single dose, 1 day), at least 5 days washout, Fluticasone Propionate Drug formulation 1 (500mcg single dose, 1 day), at least 5 days washout, Fluticasone Propionate Drug formulation 3* (500mcg single dose, 1 day), at least 5 days washout, Fluticasone Propionate Drug formulation 2 (500mcg single dose, 1 day)
  See Formulation Development in Detailed Description for details regarding differences in formulations.
  *(The asterisk) A different set of capsules from the same batch of formulation 3 is given to the subject to assess the within-subject variability and to ensure that the study is sufficiently powered to show bioequivalence between two replicates of the same formulation.
- Fluticasone Propionate Formulation Sequence 3*321: Fluticasone Propionate Formulation Sequence 3*321
  Fluticasone Propionate Drug formulation 3* (500mcg single dose, 1 day), at least 5 days washout, Fluticasone Propionate Drug formulation 3 (500mcg single dose, 1 day), at least 5 days washout, Fluticasone Propionate Drug formulation 2 (500mcg single dose, 1 day), at least 5 days washout, Fluticasone Propionate Drug formulation 1 (500mcg single dose, 1 day)
  See Formulation Development in Detailed Description for details regarding differences in formulations.
  *(The asterisk) A different set of capsules from the same batch of formulation 3 is given to the subject to assess the within-subject variability and to ensure that the study is sufficiently powered to show bioequivalence between two replicates of the same formulation.
Period: Period 1
Arm/Group | Fluticasone Propionate Formulation Sequence 1233* | Fluticasone Propionate Formulation Sequence 23*13 | Fluticasone Propionate Formulation Sequence 313*2 | Fluticasone Propionate Formulation Sequence 3*321
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Fluticasone Propionate Formulation Sequence 1233* | Fluticasone Propionate Formulation Sequence 23*13 | Fluticasone Propionate Formulation Sequence 313*2 | Fluticasone Propionate Formulation Sequence 3*321
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Fluticasone Propionate Formulation Sequence 1233* | Fluticasone Propionate Formulation Sequence 23*13 | Fluticasone Propionate Formulation Sequence 313*2 | Fluticasone Propionate Formulation Sequence 3*321
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Fluticasone Propionate Formulation Sequence 1233* | Fluticasone Propionate Formulation Sequence 23*13 | Fluticasone Propionate Formulation Sequence 313*2 | Fluticasone Propionate Formulation Sequence 3*321
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fluticasone Propionate Formulation Dequence 23*13: Fluticasone Propionate Drug formulation 2 (500mcg single dose, 1 day), at least 5 days washout, Fluticasone Propionate Drug formulation 3* (500mcg single dose, 1 day), at least 5 days washout, Fluticasone Propionate Drug formulation 1 (500mcg single dose, 1 day), at least 5 days washout, Fluticasone Propionate Drug formulation 3 (500mcg single dose, 1 day)
  See Formulation Development in Detailed Description for details regarding differences in formulations.
  *(The asterisk) A different set of capsules from the same batch of formulation 3 is given to the subject to assess the within-subject variability and to ensure that the study is sufficiently powered to show bioequivalence between two replicates of the same formulation.
- Fluticasone Propionate Formulation Sequence 3*321: Fluticasone Propionate Drug formulation 3* (500mcg single dose, 1 day), at least 5 days washout, Fluticasone Propionate Drug formulation 3 (500mcg single dose, 1 day), at least 5 days washout, Fluticasone Propionate Drug formulation 2 (500mcg single dose, 1 day), at least 5 days washout, Fluticasone Propionate Drug formulation 1 (500mcg single dose, 1 day)
  See Formulation Development in Detailed Description for details regarding differences in formulations.
  *(The asterisk) A different set of capsules from the same batch of formulation 3 is given to the subject to assess the within-subject variability and to ensure that the study is sufficiently powered to show bioequivalence between two replicates of the same formulation.
- Total: Total of all reporting groups
Arm/Group | Fluticasone Propionate Formulation Sequence 1233* | Fluticasone Propionate Formulation Dequence 23*13 | Fluticasone Propionate Formulation Sequence 313*2 | Fluticasone Propionate Formulation Sequence 3*321 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Full Range); unit: years] | 22.17 [19 to 27] | 21.67 [20 to 26] | 20.67 [19 to 23] | 26.33 [18 to 48] | 22.71 [18 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 3 | 2 | 13
  Male | 2 | 2 | 3 | 4 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 4 | 2 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 2 | 3 | 11
  White | 1 | 0 | 2 | 2 | 5
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 24
Weight (kg) [Mean (Full Range); unit: kg] | 62.6 [57.5 to 71.7] | 61.6 [50.2 to 71.7] | 64.6 [56 to 71.4] | 69.5 [57.8 to 75.1] | 64.7 [50.2 to 75.1]
Height (cm) [Mean (Full Range); unit: cm] | 169.0 [155.1 to 180.0] | 164.5 [157.8 to 169.6] | 162.7 [155.6 to 174.7] | 172.2 [163.7 to 179.1] | 167.1 [155.1 to 180.0]
BMI [Mean (Full Range); unit: kg/m2] | 22.00 [18.56 to 24.53] | 22.87 [18.82 to 28.79] | 24.4 [23.1 to 25.9] | 23.4 [19.9 to 27.3] | 23.17 [18.56 to 28.79]
FEV1 (L) [Mean (Full Range); unit: L/s] | 3.48 [2.45 to 4.20] | 3.14 [2.88 to 3.42] | 3.28 [2.47 to 4.15] | 3.97 [3.22 to 4.36] | 3.47 [2.45 to 4.36]
FEV1/FVC [Mean (Full Range); unit: ratio] | 0.892 [0.86 to 0.92] | 0.853 [0.81 to 0.91] | 0.862 [0.83 to 0.89] | 0.875 [0.84 to 0.93] | 0.870 [0.81 to 0.93]

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 the Last Quantifiable Concentration (AUC0-last) With Dose Normalization
Description: Area under the plasma concentration versus time curve from time zero (pre-dose) to the last quantifiable concentration after pulmonary dose (estimated from anatomical throats) normalization; measured as picograms multiplied by hours divided by milliliters (pg*h/mL).
Time Frame: Day 1 of Periods 1, 2, 3, and 4: pre-dose (15 minutes prior to the dosing), and 5, 10, 15, 20, 30, 45, 60 minutes, 1.5, 2, 3, 4, 6, 8, 10, 12, 14 and 24 hours (+/- 1 hour) post-dose
Population: Pharmacokinetic parameter analysis (PK) population: all participants were randomized and treated and had at least 1 of the PK parameters of primary interest in at least 1 treatment period. N=number of participants contributing to the mean.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: pg.h/mL
Groups:
- Fluticasone Propionate Formulation 1 (A-4.5 µm): Fluticasone Propionate dry powder inhaler formulation 1 (A-4.5 µm) administered via Plastiape Monodose Dry powder Inhaler on Day 1 of study period, 500mcg single dose (administered as 5 capsules and each capsule was inhaled at least two times).
- Fluticasone Propionate Formulation 2 (B-3.8 µm): Fluticasone Propionate dry powder inhaler formulation 2 (B-3.8 µm) administered via Plastiape Monodose Dry powder Inhaler on Day 1 of study period, 500mcg single dose (administered as 5 capsules and each capsule was inhaled at least two times).
- Fluticasone Propionate Formulation 3 (C-3.7 µm): Fluticasone Propionate dry powder inhaler formulation 3 (C-3.7 µm) administered via Plastiape Monodose Dry powder Inhaler on Day 1 of study period, 500mcg single dose (administered as 5 capsules and each capsule was inhaled at least two times).
- Fluticasone Propionate Formulation 3 (C-3.7 µm)*: Fluticasone Propionate dry powder inhaler formulation 3 (C-3.7 µm)* administered via Plastiape Monodose Dry powder Inhaler on Day 1 of study period, 500mcg single dose (administered as 5 capsules and each capsule was inhaled at least two times). * (The asterisk) A different set of capsules from the same batch of formulation 3 is given to the subject to assess the within-subject variability and to ensure that the study is sufficiently powered to show bioequivalence between two replicates of the same formulation.
Arm/Group | Fluticasone Propionate Formulation 1 (A-4.5 µm) | Fluticasone Propionate Formulation 2 (B-3.8 µm) | Fluticasone Propionate Formulation 3 (C-3.7 µm) | Fluticasone Propionate Formulation 3 (C-3.7 µm)*
Number analyzed (Participants) | 24 | 24 | 24 | 24
pg.h/mL | 658 [585 to 740] | 700 [622 to 787] | 716 [636 to 805] | 748 [665 to 841]
Statistical Analysis 1: Comparison: Fluticasone Propionate Formulation 1 (A-4.5 µm) vs Fluticasone Propionate Formulation 2 (B-3.8 µm); Test: Fluticasone Propionate Formulation 2 (B-3.8 µm); Reference: Fluticasone Propionate Formulation 1 (A-4.5 µm); Natural log transformed AUC0-last: mixed models analysis with sequence, period, treatment as fixed effects and subject within sequence as a random effect. All reported p-values are Bonferroni adjusted p-values; Test type: Equivalence — Bioequivalence of the two treatments was to be concluded if the 90% CIs for the ratio of geometric means for AUC0-last fell completely within (80%, 125%); p = 0.4132, Mixed Models Analysis — The threshold for statistical significane was p=0.05; ratio (%) of geometric means = 106, 90% CI 2-sided [99 to 114] — Mean difference and the 90% CI for the difference were exponentiated to provide an estimate of the ratio of adjusted geometric means (test/reference)
Statistical Analysis 2: Comparison: Fluticasone Propionate Formulation 1 (A-4.5 µm) vs Fluticasone Propionate Formulation 3 (C-3.7 µm); Test: Fluticasone Propionate Formulation 3 (C-3.7 µm); Reference: Fluticasone Propionate Formulation 1 (A-4.5 µm); Natural log transformed AUC0-last: mixed models analysis with sequence, period, treatment as fixed effects and subject within sequence as a random effect. All reported p-values are Bonferroni adjusted p-values; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.1295, Mixed Models Analysis — The threshold for statistical significane was p=0.05; ratio (%) of geometric means = 109, 90% CI 2-sided [102 to 116] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Fluticasone Propionate Formulation 1 (A-4.5 µm) vs Fluticasone Propionate Formulation 3 (C-3.7 µm)*; Test: Fluticasone Propionate Formulation 3 (C-3.7 µm)*; Reference: Fluticasone Propionate Formulation 1 (A-4.5 µm); Natural log transformed AUC0-last: mixed models analysis with sequence, period, treatment as fixed effects and subject within sequence as a random effect. All reported p-values are Bonferroni adjusted p-values; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0078, Mixed Models Analysis — The threshold for statistical significane was p=0.05; ratio (%) of geometric means = 114, 90% CI 2-sided [106 to 122] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) With Dose Normalization
Description: Cmax measured as picograms divided by milliliters (pg/mL) after pulmonary dose (estimated from anatomical throats) normalization.
Time Frame: as for outcome 1
Population: PK population; N=number of participants contributing to the mean.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Fluticasone Propionate Formulation 1 (A-4.5 µm) | Fluticasone Propionate Formulation 2 (B-3.8 µm) | Fluticasone Propionate Formulation 3 (C-3.7 µm) | Fluticasone Propionate Formulation 3 (C-3.7 µm)*
Number analyzed (Participants) | 24 | 24 | 24 | 24
pg/mL | 119 [100 to 143] | 217 [182 to 260] | 227 [190 to 271] | 254 [213 to 304]
Statistical Analysis 1: Comparison: Fluticasone Propionate Formulation 1 (A-4.5 µm) vs Fluticasone Propionate Formulation 2 (B-3.8 µm); Test: Fluticasone Propionate Formulation 2 (B-3.8 µm); Reference: Fluticasone Propionate Formulation 1 (A-4.5 µm); Natural log transformed Cmax: mixed models analysis with sequence, period, treatment as fixed effects and subject within sequence as a random effect. All reported p-values are Bonferroni adjusted p-values; Test type: Equivalence — Bioequivalence of the two treatments was to be concluded if the 90% CIs for the ratio of geometric means for Cmax fell completely within (80%, 125%); p < 0.001, Mixed Models Analysis — The threshold for statistical significane was p=0.05; ratio (%) of geometric means = 182, 90% CI 2-sided [159 to 208] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Fluticasone Propionate Formulation 1 (A-4.5 µm) vs Fluticasone Propionate Formulation 3 (C-3.7 µm); Test: Fluticasone Propionate Formulation 3 (C-3.7 µm); Reference: Fluticasone Propionate Formulation 1 (A-4.5 µm); Natural log transformed Cmax: mixed models analysis with sequence, period, treatment as fixed effects and subject within sequence as a random effect. All reported p-values are Bonferroni adjusted p-values; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.001, Mixed Models Analysis — The threshold for statistical significance was p=0.05; ratio (%) of geometric means = 190, 90% CI 2-sided [166 to 217] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Fluticasone Propionate Formulation 1 (A-4.5 µm) vs Fluticasone Propionate Formulation 3 (C-3.7 µm)*; Test: Fluticasone Propionate Formulation 3 (C-3.7 µm)*; Reference: Fluticasone Propionate Formulation 1 (A-4.5 µm); Natural log transformed Cmax: mixed models analysis with sequence, period, treatment as fixed effects and subject within sequence as a random effect. All reported p-values are Bonferroni adjusted p-values; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.001, Mixed Models Analysis — The threshold for statistical significance was p=0.05; ratio (%) of geometric means = 213, 90% CI 2-sided [186 to 244] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Description: Tmax measured as hours (h).
Time Frame: as for outcome 1
Population: PK population; N=number of participants contributing to the mean.
Measure: Median (Full Range); unit: h
Arm/Group | Fluticasone Propionate Formulation 1 (A-4.5 µm) | Fluticasone Propionate Formulation 2 (B-3.8 µm) | Fluticasone Propionate Formulation 3 (C-3.7 µm) | Fluticasone Propionate Formulation 3 (C-3.7 µm)*
Number analyzed (Participants) | 24 | 24 | 24 | 24
h | 0.51 [0.18 to 1.60] | 0.33 [0.17 to 1.10] | 0.30 [0.17 to 1.08] | 0.27 [0.17 to 1.10]

4. Secondary Outcome: Mean Residence Time (MRT)
Description: MRT measured as hours (h)
Time Frame: as for outcome 1
Population: PK population; N=number of participants contributing to the mean.
Measure: Median (Full Range); unit: h
Arm/Group | Fluticasone Propionate Formulation 1 (A-4.5 µm) | Fluticasone Propionate Formulation 2 (B-3.8 µm) | Fluticasone Propionate Formulation 3 (C-3.7 µm) | Fluticasone Propionate Formulation 3 (C-3.7 µm)*
Number analyzed (Participants) | 24 | 24 | 24 | 24
h | 11.6 [6.46 to 18.1] | 9.47 [7.07 to 13.7] | 9.41 [6.23 to 13.7] | 9.49 [6.28 to 16.5]

5. Secondary Outcome: Elimination Half Life (t1/2)
Description: t1/2 measured as hours (h)
Time Frame: as for outcome 1
Population: PK population; N=number of participants contributing to the mean.
Measure: Median (Full Range); unit: h
Arm/Group | Fluticasone Propionate Formulation 1 (A-4.5 µm) | Fluticasone Propionate Formulation 2 (B-3.8 µm) | Fluticasone Propionate Formulation 3 (C-3.7 µm) | Fluticasone Propionate Formulation 3 (C-3.7 µm)*
Number analyzed (Participants) | 24 | 24 | 24 | 24
h | 10.3 [5.74 to 17.6] | 10.3 [6.88 to 13.4] | 9.75 [6.33 to 15.6] | 10.1 [6.74 to 19.9]

ADVERSE EVENTS:
Time Frame: The duration of study participants is up to 2 months.
Groups:
- Fluticasone Propionate Formulation 1: Fluticasone Propionate Drug formulation 1 administered via Plastiape Monodose Dry powder Inhaler , 500mcg single dose.
  See Formulation Development in Detailed Description for details regarding differences in formulations
  Fluticasone Propionate Formulation 1: Fluticasone Propionate dry powder inhaler Formulation 1
  Fluticasone Propionate Formulation 2: Fluticasone Propionate dry powder inhaler Formulation 2
  Fluticasone Propionate Formulation 3: Fluticasone Propionate dry powder inhaler Formulation 3
  Fluticasone Propionate Formulation 3*: Fluticasone Propionate dry powder inhaler Formulation 3*
  *(The asterisk) A different set of capsules from the same batch of formulation 3 is given to the subject to assess the within-subject variability and to ensure that the study is sufficiently powered to show bioequivalence between two replicates of the same formulation.
- Fluticasone Propionate Formulation 2: Fluticasone Propionate Drug formulation 2 administered via Plastiape Monodose Dry powder Inhaler , 500mcg single dose.
  See Formulation Development in Detailed Description for details regarding differences in formulations
  Fluticasone Propionate Formulation 1: Fluticasone Propionate dry powder inhaler Formulation 1
  Fluticasone Propionate Formulation 2: Fluticasone Propionate dry powder inhaler Formulation 2
  Fluticasone Propionate Formulation 3: Fluticasone Propionate dry powder inhaler Formulation 3
  Fluticasone Propionate Formulation 3*: Fluticasone Propionate dry powder inhaler Formulation 3*
  *(The asterisk) A different set of capsules from the same batch of formulation 3 is given to the subject to assess the within-subject variability and to ensure that the study is sufficiently powered to show bioequivalence between two replicates of the same formulation.
- Fluticasone Propionate Formulation 3: Fluticasone Propionate Drug formulation 3 administered via Plastiape Monodose Dry powder Inhaler , 500mcg single dose.
  See Formulation Development in Detailed Description for details regarding differences in formulations
  Fluticasone Propionate Formulation 1: Fluticasone Propionate dry powder inhaler Formulation 1
  Fluticasone Propionate Formulation 2: Fluticasone Propionate dry powder inhaler Formulation 2
  Fluticasone Propionate Formulation 3: Fluticasone Propionate dry powder inhaler Formulation 3
  Fluticasone Propionate Formulation 3*: Fluticasone Propionate dry powder inhaler Formulation 3*
  *(The asterisk) A different set of capsules from the same batch of formulation 3 is given to the subject to assess the within-subject variability and to ensure that the study is sufficiently powered to show bioequivalence between two replicates of the same formulation.
- Fluticasone Propionate Formulation 3*: Fluticasone Propionate Drug formulation 3 administered via Plastiape Monodose Dry powder Inhaler , 500mcg single dose. *
  Fluticasone Propionate Formulation 1: Fluticasone Propionate dry powder inhaler Formulation 1
  Fluticasone Propionate Formulation 2: Fluticasone Propionate dry powder inhaler Formulation 2
  Fluticasone Propionate Formulation 3: Fluticasone Propionate dry powder inhaler Formulation 3
  Fluticasone Propionate Formulation 3*: Fluticasone Propionate dry powder inhaler Formulation 3*
  *(The asterisk) A different set of capsules from the same batch of formulation 3 is given to the subject to assess the within-subject variability and to ensure that the study is sufficiently powered to show bioequivalence between two replicates of the same formulation.
Arm/Group | Fluticasone Propionate Formulation 1 | Fluticasone Propionate Formulation 2 | Fluticasone Propionate Formulation 3 | Fluticasone Propionate Formulation 3*
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 4/24 | 5/24 | 5/24 | 2/24
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluticasone Propionate Formulation 1 (N=24) | Fluticasone Propionate Formulation 2 (N=24) | Fluticasone Propionate Formulation 3 (N=24) | Fluticasone Propionate Formulation 3* (N=24)
Dry Throat (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Menstrual Cramps/Pain (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Running Nose/Dry Cough (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chest Discomfort (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Funny taste (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injuries after fall/accident (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) — after Fall
Dizziness/ Lightheadedness (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin redness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-03-05): https://cdn.clinicaltrials.gov/large-docs/92/NCT01966692/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/92/NCT01966692/SAP_001.pdf